CLINICAL TRIAL: NCT03155178
Title: 96-hour Antimicrobial Persistence Assessment Following Exposure to Saline and Blotting
Brief Title: In Vivo Preoperative Skin Preparation Persistence Evaluation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EM-013953
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Results first posted 2020-02-28 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Bacterial Recovery of Skin Flora Post-product Application
MeSH Terms: interventions — chlorhexidine gluconate; 2-Propanol; Chlorhexidine; Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 3M CHG/IPA Prep (Experimental): Apply topically for 30 seconds (abdominal site) or 2 minutes (inguinal site), and allow to dry for 3 minutes.
  Interventions: Drug: 3M CHG/IPA Prep
- ChloraPrep (Active Comparator): Apply topically for 30 seconds (abdominal site) or 2 minutes (inguinal site), and allow to dry for 3 minutes.
  Interventions: Drug: ChloraPrep

INTERVENTIONS:
Drug: 3M CHG/IPA Prep — Apply topically to intact dry skin (abdominal site) for 30 seconds or moist skin (inguinal site) for 2 minutes.
  Other Names: Chlorhexidine Gluconate and Isopropyl Alcohol; CHG/IPA
  Arms: 3M CHG/IPA Prep
Drug: ChloraPrep — Apply topically to intact dry skin (abdominal site) for 30 seconds or moist skin (inguinal site) for 2 minutes.
  Other Names: Chlorhexidine Gluconate and Isopropyl Alcohol; Chlorhexidine 2% / Isopropyl alcohol 70%; CHG/IPA; ChloraPrep One-Step
  Arms: ChloraPrep

SUMMARY:
Evaluate persistent antimicrobial effectiveness of chlorhexidine gluconate containing products on abdominal and inguinal sites following a saline and wipe challenge.

DETAILED DESCRIPTION:
Persistent antimicrobial effectiveness was evaluated by measuring the regrowth of normal skin flora at 48 hours, 72 hours and 96 hours, and the suppression of regrowth relative to post-prep (10-min) at 48 hours, 72 hours and 96 hours.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any race
* Subjects in good health
* Minimum skin flora baseline requirements on abdomen and groin

Exclusion Criteria:

* Any tattoos, scars, breaks in the skin, or any form of dermatitis, or other skin disorders (including acne) on the applicable test area
* Topical antimicrobial exposure within 14 days prior to screening and treatment days
* Use of systemic or topical antibiotics, steroid medications, or any other products known to affect the normal microbial flora of the skin within 14 days prior to screening and treatment days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rozalia Olsavszky, MD, Principal Investigator — Evic / Eurofins

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a randomized, paired-comparisons design where each subject will receive two of the planned treatments, one on the left side of body and one on the right.
  Each subject provides 2 abdomen test sites, left or right, and 2 inguen test sites, left or right. Therefore 69 subjects provide 276 potential test sites.
Units Other Than Participants: test sites on skin
Groups:
- 3M CHG/IPA Prep/Abdominal Region: Experimental CHG/IPA prep was randomly assigned to the left or right side of the abdominal test site
- ChloraPrep/Abdominal Region: Active comparator CHG/IPA prep was randomly assigned to the left or right side of the abdominal test sites
- 3M CHG/IPA Prep/Inguinal Region: Experimental CHG/IPA prep was randomly assigned to the left or right side of the inguinal test site
- ChloraPrep/Inguinal Region: Active comparator prep was randomly assigned to the left or right side of the inguinal test site
Period: Overall Study
Arm/Group | 3M CHG/IPA Prep/Abdominal Region | ChloraPrep/Abdominal Region | 3M CHG/IPA Prep/Inguinal Region | ChloraPrep/Inguinal Region
Started | 69; 69 test sites on skin | 69; 69 test sites on skin | 69; 69 test sites on skin | 69; 69 test sites on skin
Completed | 62; 62 test sites on skin | 62; 62 test sites on skin | 62; 62 test sites on skin | 62; 62 test sites on skin
Not Completed | 7; 7 test sites on skin | 7; 7 test sites on skin | 7; 7 test sites on skin | 7; 7 test sites on skin
Not completed — Did not meet treatment day baseline | 7 | 7 | 7 | 7

BASELINE CHARACTERISTICS:
Population: Subjects with average treatment day baseline counts of greater than or equal to 3.00 log10 CFU/cm2 bilaterally on the abdominal region and/or greater than or equal to 5.00 log10 CFU/cm2 bilaterally on the inguinal region were included in the analysis.
  69 subjects provided 276 baseline test sites (69 rt abd, 69 lt abd, 69 rt ing, 69 lt ing).
Units Other Than Participants: test sites on skin
Groups:
- 3M CHG/IPA/Abdominal Region: Investigational CHG/IPA Prep randomly assigned to the left or right abdominal region test sites
- ChloraPrep/Abdominal Region; ChloraPrep/Inguinal Region: Active marketed comparator CHG/IPA Prep randomly assigned to the left or right abdominal region test sites
- 3M CHG/IPA/Inguinal Region: Investigational CHG/IPA Prep randomly assigned to the left or right inguiinal region test sites
- Total: Total of all reporting groups
Arm/Group | 3M CHG/IPA/Abdominal Region | ChloraPrep/Abdominal Region | 3M CHG/IPA/Inguinal Region | ChloraPrep/Inguinal Region | Total
Number analyzed (Participants) | 69 | 69 | 69 | 69 | 276
Number analyzed (test sites on skin) | 69 | 69 | 69 | 69 | 276
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 62 | 62 | 62 | 62 | 248
  >=65 years | 7 | 7 | 7 | 7 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 48 | 48 | 192
  Male | 21 | 21 | 21 | 21 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 69 | 69 | 69 | 69 | 276
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 69 | 69 | 69 | 69 | 276
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Subjects meeting treatment day baseline requirement [Count of Units; unit: test sites on skin] — Treatment day baseline requirement is defined as greater than or equal to 3.00 log10 CFU/cm^2 bilaterally on the abdomen test site and/or greater than or equal to 5.00 log10 CFU/cm^2 bilaterally on the inguinal test site.
  test sites on skin | 69 | 69 | 69 | 69 | 276

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Skin Flora Recovery Post-prep Application
Description: The primary measure of persistence is the suppression of regrowth recovery relative to baseline (log10 CFU/cm^2) of skin flora at 3 defined post-treatment sampling times.
Time Frame: Baseline, 48-hours post-treatment, 72-hours post-treatment and 96-hours post-treatment
Population: The primary analysis data set used a Modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of either > or equal to 3.0 log10 CFU/cm^2 on the abdomen test site or > or equal to 5.0 log10 CFU/cm^2 on the inguinal test site.
Measure: Mean (Standard Deviation); unit: log10 CFU/cm^2
Groups:
- Experimental Prep - Abdominal Site: Following baseline sample collection participants had 3M CHG/IPA Prep applied to their abdominal test site for 30 seconds and dry for 3 minutes.
- Active Comparator Prep - Abdominal Site: Following baseline sample collection participants had ChloraPrep applied to their abdominal test site for 30 seconds and dry for 3 minutes.
- Experimental Prep - Inguinal Site: Following baseline sample collection participants had 3M CHG/IPA Prep applied to their inguinal test site for 2 minutes and dry for 3 minutes.
- Active Comparator Prep - Inguinal Site: Following baseline sample collection participants had ChloraPrep applied to their inguinal test site for 2 minutes and dry for 3 minutes.
Arm/Group | Experimental Prep - Abdominal Site | Active Comparator Prep - Abdominal Site | Experimental Prep - Inguinal Site | Active Comparator Prep - Inguinal Site
Number analyzed (Participants) | 62 | 62 | 62 | 62
log10 CFU/cm^2
  48 hour timepoint | 1.39 (1.27) | 1.15 (1.02) | 1.97 (1.19) | 1.82 (1.10)
  72 hour timepoint | 0.89 (1.11) | 0.92 (1.05) | 1.94 (1.41) | 2.13 (1.30)
  96 hour timepoint | 1.21 (1.20) | 1.17 (1.18) | 2.39 (1.48) | 2.46 (1.52)
Statistical Analysis 1: Comparison: Experimental Prep - Abdominal Site vs Active Comparator Prep - Abdominal Site; 48-hours post-treatment time point. The primary analysis dataset used a modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of greater than or equal to 3.0 log10 CFU/cm^2 on the abdomen. The null hypothesis is that there is no difference in log10 CFU /cm^2 recovery between arms at 48-hours post-treatment; Test type: Superiority; p = 0.13, Paired t-test; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.53 to 0.07], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Experimental Prep - Abdominal Site vs Active Comparator Prep - Abdominal Site; 72-hours post-treatment time point. The primary analysis dataset used a modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of greater than or equal to 3.0 log10 CFU/cm^2 on the abdomen. The null hypothesis is that there is no difference in log10 CFU /cm^2 recovery between arms at 72-hours post-treatment; Test type: Superiority; p = 0.78, Paired t-test; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.23 to 0.30], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Experimental Prep - Abdominal Site vs Active Comparator Prep - Abdominal Site; 96-hours post-treatment time point. The primary analysis dataset used a modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of greater than or equal to 3.0 log10 CFU/cm^2 on the abdomen. The null hypothesis is that there is no difference in log10 CFU /cm^2 recovery between arms at 96-hours post-treatment; Test type: Superiority; p = 0.77, Paired t-test; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.38 to 0.29], Standard Error of Mean 0.17
Statistical Analysis 4: Comparison: Experimental Prep - Inguinal Site vs Active Comparator Prep - Inguinal Site; 48-hours post-treatment time point. The primary analysis dataset used a modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of greater than or equal to 5.0 log10 CFU/cm^2 on the inguinal. The null hypothesis is that there is no difference in log10 CFU /cm^2 recovery between arms at 48-hours post-treatment; Test type: Superiority; p = 0.37, Paired t-test; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.45 to 0.17], Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: Experimental Prep - Inguinal Site vs Active Comparator Prep - Inguinal Site; 72-hours post-treatment time point. The primary analysis dataset used a modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of greater than or equal to 5.0 log10 CFU/cm^2 on the inguinal. The null hypothesis is that there is no difference in log10 CFU /cm^2 recovery between arms at 72-hours post-treatment; Test type: Superiority; p = 0.33, Paired t-test; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.20 to 0.58], Standard Error of Mean 0.20
Statistical Analysis 6: Comparison: Experimental Prep - Inguinal Site vs Active Comparator Prep - Inguinal Site; 96-hours post-treatment time point. The primary analysis dataset used a modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of greater than or equal to 5.0 log10 CFU/cm^2 on the inguinal. The null hypothesis is that there is no difference in log10 CFU /cm^2 recovery between arms at 96-hours post-treatment; Test type: Superiority; p = 0.65, Paired t-test; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.25 to 0.39], Standard Error of Mean 0.16

2. Secondary Outcome: Change in Skin Flora Relative to 10 Minutes Post-prep Application
Description: Log10 CFU/cm^2 regrowth of skin flora, relative to 10-minute post-treatment log10 CFU/cm^2, at 3 defined post-treatment sampling times.
Time Frame: 10-minute post-treatment, 48-hours post-treatment, 72-hours post-treatment and 96-hours post-treatment
Population: The secondary analysis data set used a Modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of either > or equal to 3.0 log10 CFU/cm^2 on the abdomen test site or 5.0 log10 CFU/cm^2 on the inguinal test
Measure: Mean (Standard Deviation); unit: log10 CFU/cm^2
Arm/Group | Experimental Prep - Abdominal Site | Active Comparator Prep - Abdominal Site | Experimental Prep - Inguinal Site | Active Comparator Prep - Inguinal Site
Number analyzed (Participants) | 62 | 62 | 62 | 62
log10 CFU/cm^2
  48 hour timepoint | -0.07 (1.34) | -0.26 (1.37) | 0.24 (1.42) | 0.44 (1.56)
  72 hour timepoint | -0.57 (1.16) | -0.49 (1.35) | 0.21 (1.63) | 0.75 (1.78)
  96 hour timepoint | -0.24 (1.35) | -0.25 (1.55) | 0.66 (2.04) | 1.08 (1.81)
Statistical Analysis 1: Comparison: Experimental Prep - Abdominal Site vs Active Comparator Prep - Abdominal Site; 48-hours post-treatment time point. The primary analysis dataset used a modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of greater than or equal to 3.0 log10 CFU/cm^2 on the abdomen. The null hypothesis is that there is no difference in log10 CFU /cm^2 regrowth from the 10 minute time point between arms at 48-hours post-treatment; Test type: Superiority; p = 0.38, Paired t-test; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.63 to 0.24], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Experimental Prep - Abdominal Site vs Active Comparator Prep - Abdominal Site; 72-hours post-treatment time point. The primary analysis dataset used a modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of greater than or equal to 3.0 log10 CFU/cm^2 on the abdomen. The null hypothesis is that there is no difference in log10 CFU /cm^2 regrowth from the 10 minute time point between arms at 72-hours post-treatment; Test type: Superiority; p = 0.68, Paired t-test; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.30 to 0.45], Standard Error of Mean 0.19
Statistical Analysis 3: Comparison: Experimental Prep - Abdominal Site vs Active Comparator Prep - Abdominal Site; 96-hours post-treatment time point. The primary analysis dataset used a modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of greater than or equal to 3.0 log10 CFU/cm^2 on the abdomen. The null hypothesis is that there is no difference in log10 CFU /cm^2 regrowth from the 10 minute time point between arms at 96-hours post-treatment; Test type: Superiority; p = 0.97, Paired t-test; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.47 to 0.45], Standard Error of Mean 0.23
Statistical Analysis 4: Comparison: Experimental Prep - Inguinal Site vs Active Comparator Prep - Inguinal Site; 48-hours post-treatment time point. The primary analysis dataset used a modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of greater than or equal to 5.0 log10 CFU/cm^2 on the inguinal. The null hypothesis is that there is no difference in log10 CFU /cm^2 regrowth from the 10 minute time point between arms at 48-hours post-treatment; Test type: Superiority; p = 0.40, Paired t-test; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.27 to 0.65], Standard Error of Mean 0.23
Statistical Analysis 5: Comparison: Experimental Prep - Inguinal Site vs Active Comparator Prep - Inguinal Site; 72-hours post-treatment time point. The primary analysis dataset used a modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of greater than or equal to 5.0 log10 CFU/cm^2 on the inguinal. The null hypothesis is that there is no difference in log10 CFU /cm^2 regrowth from the 10 minute time point between arms at 72-hours post-treatment; Test type: Superiority; p = 0.03, Paired t-test — Using a Hochberg Step-up procedure the critical p value is 0.17; Mean Difference (Final Values) = 0.54, 95% CI 2-sided [0.05 to 1.03], Standard Error of Mean 0.25
Statistical Analysis 6: Comparison: Experimental Prep - Inguinal Site vs Active Comparator Prep - Inguinal Site; 96-hours post-treatment time point. The primary analysis dataset used a modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of greater than or equal to 5.0 log10 CFU/cm^2 on the inguinal. The null hypothesis is that there is no difference in log10 CFU /cm^2 regrowth from the 10 minute time point between arms at 96-hours post-treatment; Test type: Superiority; p = 0.07, Paired t-test; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-0.03 to 0.87], Standard Error of Mean 0.23

3. Other Pre Specified Outcome: Safety Outcome Evaluated by Skin Irritation (Dryness, Edema, Erythema, Rash) Assessment
Description: Skin irritation (dryness, edema, erythema, rash) assessed on the test sites using a 0-3 rating scale: 0=no reaction, 1=mild, 2=moderate, 3=severe.
Time Frame: Assessed at baseline (pre-treatment) and 10 minutes post-treatment, 48 hours post-treatment, 72 hours post-treatment, 96 hours post-treatment
Population: Subjects meeting required baseline counts: greater or equal to 3.00 log10 CFU/cm^2 on the abdominal region and greater than or or equal to 5.00 log10 CFU/cm^2 on the inguinal region.
Measure: Number; unit: sites
Groups:
- 3M CHG/IPA Prep Abdominal Region: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol 70% (IPA)
- ChloraPrep CHG/IPA Abdominal Region; 3M CHG/IPA Prep Inguinal Region; ChloraPrep CHG/IPA Inguinal Region: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70%
Arm/Group | 3M CHG/IPA Prep Abdominal Region | ChloraPrep CHG/IPA Abdominal Region | 3M CHG/IPA Prep Inguinal Region | ChloraPrep CHG/IPA Inguinal Region
Number analyzed (Participants) | 62 | 62 | 62 | 62
sites
  Dryness:Baseline pre-treatment rating=0 | 62 | 62 | 62 | 62
  Dryness:10-minute post-treatment rating=0 | 62 | 62 | 62 | 62
  Dryness:48 hours post-treatment rating=0 | 62 | 62 | 62 | 62
  Dryness:72 hours post-treatment rating=0 | 62 | 62 | 62 | 62
  Dryness:96 hours post-treatment rating=0 | 62 | 62 | 62 | 62
  Edema:Baseline pre-treatment rating=0 | 62 | 62 | 62 | 62
  Edema:10 min post-treatment rating=0 | 62 | 62 | 62 | 62
  Edema:48 hours post-treatment rating=0 | 62 | 62 | 62 | 62
  Edema:72 hours post-treatment rating=0 | 62 | 62 | 62 | 62
  Edema:96 hours post-treatment rating=0 | 62 | 62 | 62 | 62
  Erythema:Baseline pre-treatment rating=0 | 62 | 62 | 62 | 62
  Erythema:10 min post-treatment rating=0 | 62 | 62 | 62 | 62
  Erythema:48 hours post-treatment rating=0 | 62 | 62 | 62 | 62
  Erythema:72 hours post-treatment rating=0 | 62 | 62 | 62 | 62
  Erythema:96 hours post-treatment rating=0 | 62 | 62 | 62 | 62
  Rash:Baseline pre-treatment rating=0 | 62 | 62 | 62 | 62
  Rash:10 min post-treatment rating=0 | 62 | 62 | 62 | 62
  Rash:48 hours post-treatment rating=0 | 62 | 62 | 62 | 62
  Rash:72 hours post-treatment rating=0 | 62 | 62 | 62 | 62
  Rash:96 hours post-treatment rating=0 | 62 | 62 | 62 | 62

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the treatment phase of the study. Product remained on each subject's skin for approximately 96 hours.
Arm/Group | 3M CHG/IPA Prep Abdominal Region | ChloraPrep CHG/IPA Abdominal Region | 3M CHG/IPA Prep Inguinal Region | ChloraPrep CHG/IPA Inguinal Region
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/69 | 0/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/69 | 0/69 | 0/69
Other Adverse Events (participants affected / at risk) | 0/69 | 0/69 | 0/69 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT03155178/Prot_SAP_000.pdf